CLINICAL TRIAL: NCT03172975
Title: Phase 2 Study to Assess the Safety, Efficacy and Immunogenicity of Na-GST-1/Alhydrogel Co-administered With Different Toll-Like Receptor Agonists in Hookworm- Naïve Adults
Brief Title: Efficacy of Na-GST-1/Alhydrogel Hookworm Vaccine Assessed by Controlled Challenge Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: George Washington University (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Maria Elena Bottazzi PhD, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-38292; U01AI129789 (NIH)
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Hookworm Infections
Keywords: Controlled infection; Na-GST-1; Hookworm vaccine
MeSH Terms: conditions — Hookworm Infections | interventions — Albendazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants and investigators will be blinded to study product allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Na-GST-1/Alhydrogel (Experimental): 100 µg Na-GST-1/Alhydrogel administered intramuscularly in the deltoid on study days 0, 56 and 112 followed by controlled human hookworm infection with 50 infectious Necator americanus larvae on study day 140.
  Interventions: Biological: Na-GST-1/Alhydrogel; Drug: Albendazole; Other: Necator americanus Larval Inoculum
- Na-GST-1/Alhydrogel + CPG 10104 (Experimental): 100 µg Na-GST-1/Alhydrogel co-administered with 500 µg CPG 10104 delivered intramuscularly in the deltoid on study days 0, 56 and 112 followed by controlled human hookworm infection with 50 infectious Necator americanus larvae on study day 140.
  Interventions: Biological: Na-GST-1/Alhydrogel + CPG 10104; Drug: Albendazole; Other: Necator americanus Larval Inoculum
- Na-GST-1/Alhydrogel + GLA-AF (Experimental): 100 µg Na-GST-1/Alhydrogel co-administered with 5 µg GLA-AF delivered intramuscularly in the deltoid on study days 0, 56 and 112 followed by controlled human hookworm infection with 50 infectious Necator americanus larvae on study day 140.
  Interventions: Biological: Na-GST-1/Alhydrogel + GLA-AF; Drug: Albendazole; Other: Necator americanus Larval Inoculum
- Saline Placebo (Placebo Comparator): Sterile saline placebo delivered intramuscularly in the deltoid on study days 0, 56 and 112 followed by controlled human hookworm infection with 50 infectious Necator americanus larvae on study day 140.
  Interventions: Biological: Placebo; Drug: Albendazole; Other: Necator americanus Larval Inoculum

INTERVENTIONS:
Biological: Na-GST-1/Alhydrogel — Recombinant Necator americanus Glutathione-S Transferase adjuvanted with Alhydrogel
  Other Names: Necator americanus Glutathione-S Transferase
  Arms: Na-GST-1/Alhydrogel
Biological: Na-GST-1/Alhydrogel + CPG 10104 — Recombinant Necator americanus Glutathione-S Transferase adjuvanted with Alhydrogel and co-administered with CPG 10104, a synthetic oligodeoxynucleotide
  Arms: Na-GST-1/Alhydrogel + CPG 10104
Biological: Na-GST-1/Alhydrogel + GLA-AF — Recombinant Necator americanus Glutathione-S Transferase adjuvanted with Alhydrogel and co-administered with an aqueous formulation of Glucopyranosyl-Lipid A (GLA-AF)
  Arms: Na-GST-1/Alhydrogel + GLA-AF
Biological: Placebo — Physiological sterile saline solution
  Arms: Saline Placebo
Drug: Albendazole — Treatment with 3 daily oral doses of 400 mg albendazole at end of study.
Other: Necator americanus Larval Inoculum — 50 infectious Necator americanus larvae applied via dermal application (challenge infection).

SUMMARY:
This study evaluates the efficacy, safety and immunogenicity of different formulations of the Na-GST-1 hookworm vaccine using a controlled human hookworm infection model in healthy, hookworm-naive adults.

DETAILED DESCRIPTION:
Double blind, randomized, controlled, Phase 2 clinical trial in hookworm-unexposed adults living in the metropolitan area of Washington, DC. Subjects will receive three doses of the assigned vaccine formulation, or saline placebo, delivered intramuscularly on approximately Days 0, 56, and 112.

Subjects will be challenged with 50 infectious N. americanus larvae 4 weeks after 3rd vaccination. Fecal samples will be collected weekly starting 4 weeks post-challenge. Albendazole will be administered 20 weeks post-challenge to cure infections. Subjects will be followed until 10 months after their final vaccination.

Safety of vaccination will be measured from the time of each study vaccination (Day 0) through 14 days after each study vaccination by the occurrence of solicited injection site and systemic reactogenicity events. Safety of CHHI will be measure from the time of larval application (Day 140) through the first day of treatment with albendazole (Day 280).

Unsolicited non-serious adverse events (AEs) will be collected until approximately 1 month following each study vaccination and from study Day 140 (day of CHHI) through Day 280.

New-onset chronic medical conditions and Serious Adverse Events (SAEs) will be collected from the time of the first study vaccination through approximately 10 months after the third study vaccination (final visit). Clinical laboratory evaluations for safety will be performed on venous blood collected approximately 14 days after each vaccination and CHHI.

Immunogenicity testing will include IgG antibody responses to Na-GST-1, by a qualified indirect enzyme-linked immunosorbent assay (ELISA), on serum obtained prior to each study vaccination and CHHI, and at time points after each vaccination and after CHHI (see Appendix A); the affinity of vaccine-induced antibodies against Na-GST-1 using Surface Plasmon Resonance; the functional activity of vaccine-induced antibodies via in vitro enzyme neutralization assay; antigen-specific memory B cell responses; and, the innate immune responses to each of the TLR receptor immunostimulants.

Parasitological testing will include microscopic fecal egg detection by a qualified saline flotation technique, fecal egg counts by the McMaster method, fecal PCR for hookworm DNA, and peripheral eosinophil counts.

Recruitment and enrollment into the study will occur on an ongoing basis, with each group being recruited and vaccinated in sequence.

48 subjects will be enrolled into 4 groups of 12. Subjects will be enrolled sequentially and upon enrollment will be randomized to one of the following IP assignments in a double-blind fashion:

* Group 1 IP allocation (n=12 subjects): 12 subjects will receive 100µg Na-GST-1/Alhydrogel® delivered by IM injection in the deltoid muscle.
* Group 2 IP allocation (n=12): 12 subjects will receive Na-GST-1/Alhydrogel® plus 500µg CpG 10104 delivered by IM injection in the deltoid muscle.
* Group 3 IP allocation (n=12): 12 subjects will receive Na-GST-1/Alhydrogel® plus 5µg GLA-AF delivered by IM injection in the deltoid muscle.
* Group 4 IP allocation (n=12): 12 subjects will receive sterile saline delivered by IM injection in the deltoid muscle.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant females between 18 and 45 years, inclusive.
2. Good general health as determined by means of the screening procedures1.
3. Available for the duration of individual subject study participation (14 months).
4. Willingness to participate in the study as evidenced by signing the informed consent document.
5. Able to understand and comply with planned study procedures.

Exclusion Criteria:

1. Pregnancy as determined by a positive urine human choriogonadotropin (hCG) test (if female).
2. Subject unwilling to use effective contraception for a minimum of 30 days prior to vaccination and up until documentation of clearance of hookworm infection post-CHHI (if female and not surgically sterile, abstinent from intercourse with a male partner, in a monogamous relationship with a vasectomized partner, at least 2 years post-menopausal, or determined otherwise by medical evaluation to be sterile).
3. Currently lactating and breast-feeding or plans to breastfeed at any given time from the first study vaccination until clearance of hookworm infection post-CHHI (if female).
4. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, gastrointestinal, diabetes, or renal disease by history, physical examination, and/or laboratory studies.
5. Has a diagnosis of schizophrenia, bipolar disease or other major psychiatric condition that would make compliance with study visits/procedures difficult (e.g., subject with psychoses or history of suicide attempt or gesture in the 3 years before study entry, ongoing risk for suicide).
6. Known or suspected immunodeficiency or immunosuppression as a result of an underlying illness or treatment (causes for immunosuppression may include, but are not limited to, poorly-controlled diabetes mellitus, chronic liver disease, renal insufficiency, active neoplastic disease or a history of hematologic malignancy, connective tissue disease, organ transplant).
7. Laboratory evidence of liver disease (alanine aminotransferase [ALT] greater than 1.25-times the upper reference limit).
8. Laboratory evidence of renal disease (serum creatinine greater than 1.25-times the upper reference limit, or urine dipstick testing positive for glucose or more than trace protein).
9. Laboratory evidence of hematologic disease (hemoglobin <11.1 g/dl [females] or <12.5 g/dl [males]; absolute leukocyte count <3400/mm3 or >10.8 x 103/mm3; absolute eosinophil count <500/mm3; or platelet count <140,000/mm3).
10. Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.
11. Planned participation in another investigational vaccine or drug trial within 30 days of starting this study or until the last study visit (this may include other licensed or unlicensed vaccines, drugs, biologics, devices, blood products, or medications).
12. Volunteer has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 24 months.
13. Positive fecal occult blood test at screening.
14. Infection with a pathogenic intestinal helminth as determined by stool examination for ova and parasites at screening.
15. History of iron deficiency anemia or laboratory evidence of iron deficiency (serum ferritin concentration below the lower reference limit).
16. History of hypoalbuminemia.
17. History of a severe allergic reaction or anaphylaxis.
18. Severe asthma as defined by the need for daily use of inhalers, or emergency clinic visit or hospitalization within 6 months of the volunteer's expected first vaccination in the study.
19. Positive test for hepatitis B surface antigen (HBsAg).
20. Positive confirmatory test for HIV infection.
21. Positive confirmatory test for hepatitis C virus (HCV) infection.
22. Using or intends to continue using oral or parenteral corticosteroids, high-dose inhaled corticosteroids (>800 μg/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs within 30 days of the volunteer's expected first vaccination in this study or planned use during the study.
23. Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to the volunteer's expected first vaccination in the study.
24. Receipt of immunoglobin or other blood products (with exception of Rho D immunoglobulin) within 90 days of the planned first study vaccination.
25. Known allergy to albendazole, amphotericin B or gentamicin.
26. History of previous infection with hookworm or continuous residence for more than 6 months in a community where hookworm is endemic.
27. Current or past scars, tattoos, or other disruptions of skin integrity at the intended site of larval application.
28. Previous receipt of the Na-GST-1/Alhydrogel® hookworm vaccine.
29. History of a surgical splenectomy.
30. Pre-existing autoimmune or antibody-mediated diseases including but not limited to: systemic lupus erythematosis, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia; or laboratory evidence of possible autoimmune disease determined by a positive anti-dsDNA titer, positive rheumatoid factor, and/or proteinuria (greater than trace protein on urine dipstick testing).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Diemert, MD, Principal Investigator — George Washington University
Locations (1):
- George Washington University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
GW provided agreement with that NIAID that it will make publicly available all final research data resulting from this U01 clinical trial, in a timely fashion following closure of the clinical trial (not more than 12 months after the last subject follow-up visit). At no time will subject identifying information be made publically available.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Within 12 months of final study visit.
Access Criteria: To be determined.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and enrollment occurred on an ongoing basis, with each group being recruited and vaccinated in parallel. Participants were enrolled sequentially and upon enrollment were randomized to one of the four groups.
Period: Overall Study
Arm/Group | Na-GST-1/Alhydrogel | Na-GST-1/Alhydrogel + CPG 10104 | Na-GST-1/Alhydrogel + GLA-AF | Saline Placebo
Started | 10 | 9 | 10 | 10
Completed | 9 | 5 | 10 | 8
Not Completed | 1 | 4 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Na-GST-1/Alhydrogel | Na-GST-1/Alhydrogel + CPG 10104 | Na-GST-1/Alhydrogel + GLA-AF | Saline Placebo | Total
Number analyzed (Participants) | 10 | 9 | 10 | 10 | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.1 (4.6) | 30.4 (8.2) | 24.7 (3.3) | 26.1 (3.45) | 26.7 (5.4)
Age, Customized [Median (Inter-Quartile Range); unit: Years]
  Age, Continuous | 25.5 [19.0 to 34.0] | 29.0 [21.0 to 44.0] | 23.5 [21.0 to 30.0] | 25.5 [22.0 to 31.0] | 26.0 [19.0 to 44.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 6 | 7 | 22
  Male | 6 | 4 | 4 | 3 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Race: Asian | 0 | 0 | 4 | 1 | 5
  Race: Black or African American | 1 | 1 | 0 | 1 | 3
  Race: Other | 1 | 2 | 0 | 2 | 5
  Race: White | 8 | 5 | 6 | 6 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 1 | 3 | 1 | 2 | 7
  Ethnicity: Not Hispanic or Latino | 9 | 6 | 9 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Detectable Hookworm Infection
Description: Proportion of subjects with detectable hookworm eggs, at any time point, in fecal samples, as determined by microscopy using the qualified saline flotation technique
Time Frame: On Study Days 175, 182, 189, 203, 217, 231, 245, 259, 273, and 280.
Population: The number of participants analyzed each week varies due to participants missing that visit.
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: Na-GST-1/Alhydrogel: 100 µg ˆNaˆ-GST-1/Alhydrogel administered intramuscularly in the deltoid on study days 0, 56 and 112 followed by controlled human hookworm infection with 50 infectious Necator americanus larvae on study day 140.
- Group 2: Na-GST-1/Alhydrogel + CPG 10104: 100 µg ˆNaˆ-GST-1/Alhydrogel co-administered with 500 µg CPG 10104 delivered intramuscularly in the deltoid on study days 0, 56 and 112 followed by controlled human hookworm infection with 50 infectious Necator americanus larvae on study day 140.
- Group 3: Na-GST-1/Alhydrogel + GLA-AF: 100 µg ˆNaˆ-GST-1/Alhydrogel co-administered with 5 µg GLA-AF delivered intramuscularly in the deltoid on study days 0, 56 and 112 followed by controlled human hookworm infection with 50 infectious Necator americanus larvae on study day 140.
- Group 4: Saline Placebo: Sterile saline placebo delivered intramuscularly in the deltoid on study days 0, 56 and 112 followed by controlled human hookworm infection with 50 infectious Necator americanus larvae on study day 140.
Arm/Group | Group 1: Na-GST-1/Alhydrogel | Group 2: Na-GST-1/Alhydrogel + CPG 10104 | Group 3: Na-GST-1/Alhydrogel + GLA-AF | Group 4: Saline Placebo
Number analyzed (Participants) | 9 | 5 | 10 | 9
Participants
  Day 175: number analyzed (Participants) | 8 | 5 | 10 | 9
  Day 175 | 0 | 0 | 0 | 0
  Day 182: number analyzed (Participants) | 9 | 3 | 10 | 8
  Day 182 | 0 | 0 | 0 | 1
  Day 189: number analyzed (Participants) | 8 | 5 | 10 | 8
  Day 189 | 0 | 0 | 0 | 2
  Day 203: number analyzed (Participants) | 9 | 5 | 9 | 7
  Day 203 | 4 | 1 | 3 | 2
  Day 217: number analyzed (Participants) | 9 | 2 | 8 | 9
  Day 217 | 3 | 1 | 4 | 4
  Day 231: number analyzed (Participants) | 9 | 4 | 10 | 9
  Day 231 | 4 | 1 | 6 | 4
  Day 245: number analyzed (Participants) | 8 | 3 | 10 | 8
  Day 245 | 3 | 0 | 5 | 3
  Day 259: number analyzed (Participants) | 9 | 2 | 9 | 7
  Day 259 | 2 | 0 | 4 | 4
  Day 273: number analyzed (Participants) | 8 | 4 | 10 | 7
  Day 273 | 2 | 0 | 6 | 3
  Day 280: number analyzed (Participants) | 9 | 2 | 8 | 7
  Day 280 | 3 | 0 | 5 | 3

2. Primary Outcome: Incidence of Serious Adverse Events
Description: Frequency of study vaccine-related Serious Adverse Events from the time of the first study vaccination through approximately 10 months after the last study vaccination.
Time Frame: Beginning on Day 0 when the first dose is received and ending on Day 380 (final study visit).
Measure: Count of Participants; unit: Participants
Groups:
- Na-GST-1/Alhydrogel: 100 µg ˆNaˆ-GST-1/Alhydrogel administered intramuscularly in the deltoid on study days 0, 56 and 112 followed by controlled human hookworm infection with 50 infectious Necator americanus larvae on study day 140.
- Na-GST-1/Alhydrogel + CPG 10104: 100 µg ˆNaˆ-GST-1/Alhydrogel co-administered with 500 µg CPG 10104 delivered intramuscularly in the deltoid on study days 0, 56 and 112 followed by controlled human hookworm infection with 50 infectious Necator americanus larvae on study day 140.
- Na-GST-1/Alhydrogel + GLA-AF: 100 µg ˆNaˆ-GST-1/Alhydrogel co-administered with 5 µg GLA-AF delivered intramuscularly in the deltoid on study days 0, 56 and 112 followed by controlled human hookworm infection with 50 infectious Necator americanus larvae on study day 140.
Arm/Group | Na-GST-1/Alhydrogel | Na-GST-1/Alhydrogel + CPG 10104 | Na-GST-1/Alhydrogel + GLA-AF | Saline Placebo
Number analyzed (Participants) | 10 | 9 | 10 | 10
Participants | 0 | 0 | 0 | 0

3. Primary Outcome: Incidence of Solicited Injection Site and Systemic Reactogenicity
Description: Frequency of solicited injection site and systemic reactogenicity, graded by severity, on the day of each study vaccination through 14 days after each study vaccination.
Time Frame: Dose 1: Days 0, 3, 7, 14; Dose 2: Days 56, 59, 63, 70; Dose 3: Days 112, 115, 119, 126
Population: 39 participants received the first dose of the study product, 37 participants received the second dose of the study product, and 36 participants received the third and final dose of the study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Na-GST-1/Alhydrogel | Group 2: Na-GST-1/Alhydrogel + CPG 10104 | Group 3: Na-GST-1/Alhydrogel + GLA-AF | Group 4: Saline Placebo
Number analyzed (Participants) | 10 | 9 | 10 | 10
Participants
  Number of Participants Reporting Solicited Adverse Events Post Dose #1 | 10 | 9 | 10 | 7
  Number of Participants Reporting Solicited Adverse Events Post Dose #2: number analyzed (Participants) | 9 | 8 | 10 | 10
  Number of Participants Reporting Solicited Adverse Events Post Dose #2 | 9 | 7 | 9 | 5
  Number of Participants Reporting Solicited Adverse Events Post Dose #3: number analyzed (Participants) | 9 | 7 | 10 | 10
  Number of Participants Reporting Solicited Adverse Events Post Dose #3 | 8 | 7 | 9 | 7

4. Primary Outcome: Incidence of Solicited Adverse Events
Description: Frequency of solicited adverse events, graded by severity, on the day of CHHI through study Day 280
Time Frame: Day of CHHI, Day 140, and study days: 143, 147, 154, 175, 182, 189, 196, 203, 210, 217, 224, 231, 238, 245, 252, 259, 266, 273, 280. Day 280 is the day of anti-worm treatment.
Population: Number of participants reporting solicited adverse events during CHHI phase of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Na-GST-1/Alhydrogel | Na-GST-1/Alhydrogel + CPG 10104 | Na-GST-1/Alhydrogel + GLA-AF | Saline Placebo
Number analyzed (Participants) | 9 | 5 | 10 | 9
Participants | 8 | 5 | 10 | 9

5. Primary Outcome: Incidence of Clinical Safety Laboratory Abnormalities
Description: Frequency of clinical safety laboratory adverse events.
Time Frame: Study days: 0, 14, 56, 70, 112, 126, 140, 154, 175, 189, 203, 217, 231, 259, 280.
Population: 39 participants received at least 1 study vaccination and 33 participants received the CHHI.
Measure: Count of Participants; unit: Participants
Arm/Group | Na-GST-1/Alhydrogel | Na-GST-1/Alhydrogel + CPG 10104 | Na-GST-1/Alhydrogel + GLA-AF | Saline Placebo
Number analyzed (Participants) | 10 | 9 | 10 | 10
Participants
  Number of Participants reporting Clinical Laboratory Adverse Event during Vaccination Phase | 1 | 3 | 0 | 2
  Number of Participants reporting Clinical Laboratory Adverse Event during CHHI Phase: number analyzed (Participants) | 9 | 5 | 10 | 9
  Number of Participants reporting Clinical Laboratory Adverse Event during CHHI Phase | 7 | 3 | 9 | 7

6. Primary Outcome: Incidence of Unsolicited Adverse Events
Description: Frequency of unsolicited adverse events, graded by severity, from the time of each study vaccination through approximately 1 month after each study vaccination; and from the time of CHHI through treatment with albendazole (Day 280)
Time Frame: From Dose 1 on Day 0 until anti-worm treatment on Day 280.
Population: 39 participants received Dose #1, 37 participants received Dose #2, 36 participants received Dose #3, and 33 participants received the CHHI.
Measure: Count of Participants; unit: Participants
Arm/Group | Na-GST-1/Alhydrogel | Na-GST-1/Alhydrogel + CPG 10104 | Na-GST-1/Alhydrogel + GLA-AF | Saline Placebo
Number analyzed (Participants) | 10 | 9 | 10 | 10
Participants
  Participants Reporting Unsolicited AEs up to 28 Days After Dose #1 | 5 | 6 | 4 | 8
  Participants Reporting Unsolicited AEs up to 28 Days After Dose #2: number analyzed (Participants) | 9 | 8 | 10 | 10
  Participants Reporting Unsolicited AEs up to 28 Days After Dose #2 | 3 | 5 | 6 | 6
  Participants Reporting Unsolicited AEs up to 28 Days After Dose #3: number analyzed (Participants) | 9 | 7 | 10 | 10
  Participants Reporting Unsolicited AEs up to 28 Days After Dose #3 | 6 | 4 | 5 | 7
  Participants Reporting Unsolicited AEs post-CHHI: number analyzed (Participants) | 9 | 5 | 10 | 9
  Participants Reporting Unsolicited AEs post-CHHI | 9 | 5 | 10 | 9

7. Primary Outcome: Incidence of New-onset Chronic Medical Conditions
Description: Frequency of new-onset chronic medical conditions through approximately 10 months after the third study vaccination.
Time Frame: Entire duration of the study. Beginning Day 0, day of first dose, until Day 380, final study visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Na-GST-1/Alhydrogel | Na-GST-1/Alhydrogel + CPG 10104 | Na-GST-1/Alhydrogel + GLA-AF | Saline Placebo
Number analyzed (Participants) | 10 | 9 | 10 | 10
Participants | 0 | 0 | 0 | 0

8. Primary Outcome: Incidence of Adverse Events of Special Interest
Description: Frequency of Adverse Events of Special Interest through approximately 10 months after the third study vaccination.
Time Frame: Entire duration of the study. Beginning Day 0, day of first dose, until Day 380, final study visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Na-GST-1/Alhydrogel | Na-GST-1/Alhydrogel + CPG 10104 | Na-GST-1/Alhydrogel + GLA-AF | Saline Placebo
Number analyzed (Participants) | 10 | 9 | 10 | 10
Participants | 0 | 0 | 0 | 0

9. Secondary Outcome: Fecal Egg Counts
Description: Fecal egg counts as determined by microscopy using the McMaster method, weekly from Weeks 5 through 20 post-CHHI
Time Frame: Week 5 and Week 20 post-CHHI. Study days: 175, 182, 189, 203, 217, 231, 245, 259, 273, and 280.
Population: The number of participants analyzed each week varies due to participants missing that visits and/or that visit occurring too far out of window.
Measure: Mean (Standard Deviation); unit: Eggs
Arm/Group | Na-GST-1/Alhydrogel | Na-GST-1/Alhydrogel + CPG 10104 | Na-GST-1/Alhydrogel + GLA-AF | Saline Placebo
Number analyzed (Participants) | 9 | 5 | 10 | 9
Eggs
  Week 5 post-CHHI (Day 175): number analyzed (Participants) | 8 | 5 | 10 | 9
  Week 5 post-CHHI (Day 175) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Week 6 post-CHHI (Day 182): number analyzed (Participants) | 9 | 3 | 10 | 8
  Week 6 post-CHHI (Day 182) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 4.2 (11.8)
  Week 7 post-CHHI (Day 189): number analyzed (Participants) | 8 | 5 | 10 | 8
  Week 7 post-CHHI (Day 189) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 10.4 (23.5)
  Week 9 post-CHHI (Day 203): number analyzed (Participants) | 9 | 5 | 9 | 7
  Week 9 post-CHHI (Day 203) | 11.1 (16.7) | 0.0 (0.0) | 5.6 (11.8) | 31.0 (58.1)
  Week 10 post-CHHI (Day 217): number analyzed (Participants) | 9 | 2 | 8 | 9
  Week 10 post-CHHI (Day 217) | 7.4 (12.1) | 0.0 (0.0) | 22.9 (41.7) | 38.9 (62.9)
  Week 12 post-CHHI (Day 231): number analyzed (Participants) | 9 | 4 | 10 | 9
  Week 12 post-CHHI (Day 231) | 14.8 (19.4) | 0.0 (0.0) | 48.3 (88.7) | 29.6 (58.8)
  Week 14 post-CHHI (Day 245): number analyzed (Participants) | 8 | 3 | 10 | 8
  Week 14 post-CHHI (Day 245) | 16.7 (34.5) | 0.0 (0.0) | 35.0 (50.0) | 14.6 (30.1)
  Week 16 post-CHHI (Day 259): number analyzed (Participants) | 9 | 2 | 9 | 7
  Week 16 post-CHHI (Day 259) | 31.5 (72.9) | 0.0 (0.0) | 59.3 (89.8) | 31.0 (29.5)
  Week 18 post-CHHI (Day 273): number analyzed (Participants) | 8 | 4 | 10 | 7
  Week 18 post-CHHI (Day 273) | 16.7 (35.6) | 0.0 (0.0) | 33.3 (43.7) | 38.1 (48.8)
  Week 20 post-CHHI (Day 280): number analyzed (Participants) | 9 | 2 | 8 | 7
  Week 20 post-CHHI (Day 280) | 13.0 (23.2) | 0.0 (0.0) | 35.4 (52.3) | 16.7 (23.6)

10. Secondary Outcome: Anti-Na-GST-1 IgG Antibody Response
Description: Anti-Na-GST-1 IgG antibody response as measured in Arbitrary Units per milliliter (AU/mL) of serum, determined by a qualified indirect enzyme-linked immunosorbent assay (ELISA) at approximately 14 days after each vaccination, and approximately 1, 2, 4, 6, 7, 8 and 10 months after the third dose. Levels of IgG antibodies against Na-GST-1 were converted to AUs by homologous interpolation of Optical Density readings at 492nm (OD492) from a standard calibration curve derived from serial dilutions of a human standard reference serum pool collected from high IgG responders (OD492 ≥ 1.000).
Time Frame: Study days: 14, 70, 126, 140, 175, 189, 231, 280, 320, and 380
Population: The number of participants analyzed each week varies due to participants missing that visits and/or that visit occurring too far out of window. Additionally, 39 participants received Dose 1, 37 participants received Dose 2, 36 participants received Dose 3, and 33 participants received the CHHI.
Measure: Mean (Standard Deviation); unit: Arbitrary Units (AUs) per milliliter
Arm/Group | Na-GST-1/Alhydrogel | Na-GST-1/Alhydrogel + CPG 10104 | Na-GST-1/Alhydrogel + GLA-AF | Saline Placebo
Number analyzed (Participants) | 10 | 9 | 10 | 10
Arbitrary Units (AUs) per milliliter
  Day 14 | 1.7 (0.9) | 1.4 (0.0) | 1.4 (0.0) | 1.7 (1.0)
  Day 70 (14 days post Dose 2): number analyzed (Participants) | 8 | 7 | 10 | 9
  Day 70 (14 days post Dose 2) | 5.6 (1.1) | 34.8 (30.9) | 26.7 (65.5) | 2.0 (1.8)
  Day 126 (14 days post Dose 3): number analyzed (Participants) | 9 | 7 | 10 | 10
  Day 126 (14 days post Dose 3) | 21.1 (32.4) | 55.3 (65.4) | 18.7 (23.3) | 1.4 (0.0)
  Day 140 (1 month post Dose 3): number analyzed (Participants) | 9 | 5 | 10 | 9
  Day 140 (1 month post Dose 3) | 8.5 (5.1) | 31.0 (29.5) | 10.9 (12.7) | 2.2 (2.3)
  Day 175 (2 months post Dose 3): number analyzed (Participants) | 9 | 6 | 10 | 9
  Day 175 (2 months post Dose 3) | 6.9 (5.2) | 42.6 (72.1) | 7.7 (7.9) | 1.7 (1.0)
  Day 189 (4 months post Dose 3): number analyzed (Participants) | 9 | 5 | 10 | 9
  Day 189 (4 months post Dose 3) | 7.1 (5.8) | 26.3 (28.4) | 6.2 (6.6) | 2.2 (2.3)
  Day 231 (6 months post Dose 3): number analyzed (Participants) | 9 | 4 | 10 | 9
  Day 231 (6 months post Dose 3) | 6.3 (4.4) | 35.1 (53.3) | 5.2 (5.8) | 2.3 (2.6)
  Day 280 (7 months post Dose 3): number analyzed (Participants) | 9 | 4 | 10 | 8
  Day 280 (7 months post Dose 3) | 4.5 (2.9) | 21.6 (26.7) | 4.0 (3.8) | 2.4 (2.6)
  Day 320 (8 months post Dose 3): number analyzed (Participants) | 9 | 5 | 10 | 8
  Day 320 (8 months post Dose 3) | 4.6 (3.0) | 22.8 (35.8) | 3.8 (3.1) | 2.6 (3.3)
  Day 380 (10 months post Dose 3): number analyzed (Participants) | 9 | 4 | 10 | 8
  Day 380 (10 months post Dose 3) | 3.9 (3.4) | 110 (11.6) | 3.1 (3.4) | 2.3 (2.3)

ADVERSE EVENTS:
Time Frame: For the Vaccination phase, solicited AEs were collected from the day of study vaccination through 14 days after each study vaccination and unsolicited AEs were collected from the day of study vaccination through 28 days after each vaccination. For the CHHI phase, solicited adverse events were collected from day of hookworm larvae administration (day 140) through day 280, the day albendazole treatment and unsolicited AEs were collected from day 140 through day 297.
Description: During vaccination phase, solicited adverse events were collected via a participant completed paper symptom diary for 14 days following each vaccination. During CHHI phase, solicited adverse events were collected via a paper participant symptom diary which participants completed daily. The vaccination phase consisted of 39 participants (Group 1: 10, Group 2: 9, Group 3: 10, Group 4: 10) and the CHHI phase consisted of 32 participants (Group 1: 9, Group 2: 5, Group 3: 10, Group 4: 9).
Arm/Group | Na-GST-1/Alhydrogel | Na-GST-1/Alhydrogel + CPG 10104 | Na-GST-1/Alhydrogel + GLA-AF | Saline Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/9 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 10/10 | 9/9 | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Na-GST-1/Alhydrogel (N=10) | Na-GST-1/Alhydrogel + CPG 10104 (N=9) | Na-GST-1/Alhydrogel + GLA-AF (N=10) | Saline Placebo (N=10)
Hospitalization (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Alcohol Intoxication
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Na-GST-1/Alhydrogel (N=10) | Na-GST-1/Alhydrogel + CPG 10104 (N=9) | Na-GST-1/Alhydrogel + GLA-AF (N=10) | Saline Placebo (N=10)
Brachycardia (Cardiac disorders) | 1 | 0 | 4 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Dry Eye (Eye disorders) | 1 | 0 | 0 | 0
Lacrimation Increased (Eye disorders) | 0 | 1 | 0 | 0
Ocular Hyperaemia (Eye disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 6
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Injection Site Bruising (General disorders) | 1 | 1 | 0 | 0
Chills (General disorders) | 0 | 2 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 3 | 3
Injection Site Haemorrhage (General disorders) | 0 | 0 | 2 | 1
Injection Site Pain (General disorders) | 0 | 0 | 0 | 1
Ear Injection (Infections and infestations) | 1 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 4 | 6
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Acrodermatitis (Infections and infestations) | 0 | 0 | 0 | 1
Oropharyngeal Gonococcal Infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 1 | 0 | 2
White Blood Cell Count Decreased (Investigations) | 1 | 0 | 0 | 1
Blood Pressure Diastolic Increased (Investigations) | 0 | 2 | 0 | 0
Eosinophil Count Increased (Investigations) | 0 | 1 | 0 | 0
White Blood Cell Count Increased (Investigations) | 0 | 1 | 0 | 0
Neutrophil Count Decreased (Investigations) | 0 | 0 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 2
Headache (Nervous system disorders) | 2 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 2 | 0
Breast Tenderness (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Premenstrual Syndrome (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 | 3 | 0 | 0
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0/9 | 0/5 | 1 | 0/9 — CHHI Phase
Brachycardia (Cardiac disorders) | 0/9 | 0/5 | 4 | 1/9 — CHHI Phase
Tachycardia (Cardiac disorders) | 0/9 | 0/5 | 1 | 2/9 — CHHI Phase
Ocular Hyperaemia (Eye disorders) | 0/9 | 0/5 | 0 | 1/9 — CHHI Phase
Abdominal Distension (Gastrointestinal disorders) | 3/9 | 0/5 | 0 | 1/9 — CHHI Phase
Abdominal Pain (Gastrointestinal disorders) | 2/9 | 0/5 | 0 | 0/9 — CHHI Phase
Flatulence (Gastrointestinal disorders) | 6/9 | 0/5 | 6 | 1/9 — CHHI Phase
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 5/9 | 0/5 | 0 | 0/9 — CHHI Phase
Nausea (Gastrointestinal disorders) | 1/9 | 0/5 | 0 | 0/9 — CHHI Phase
Toothache (Gastrointestinal disorders) | 1/9 | 0/5 | 0 | 1/9 — CHHI Phase
Constipation (Gastrointestinal disorders) | 0/9 | 1/5 | 0 | 2/9 — CHHI Phase
Apthous Ulcer (Gastrointestinal disorders) | 0/9 | 0/5 | 1 | 0/9 — CHHI Phase
Diarrhoea (Gastrointestinal disorders) | 0/9 | 0/5 | 1 | 0/9 — CHHI Phase
Application Site Discolouration (General disorders) | 8/9 | 0/5 | 7 | 6/9 — CHHI Phase
Pyrexia (General disorders) | 0/9 | 0/5 | 1 | 1/9 — CHHI Phase
Fatigue (General disorders) | 0/9 | 0/5 | 0 | 1/9 — CHHI Phase
Oedema (General disorders) | 0/9 | 0/5 | 0 | 1/9 — CHHI Phase
Bronchitis (Infections and infestations) | 1/9 | 0/5 | 0 | 1/9 — CHHI Phase
Cellulitis (Infections and infestations) | 2/9 | 0/5 | 0 | 0/9 — CHHI Phase
Upper Respiratory Tract Infection (Infections and infestations) | 2/9 | 3/5 | 5 | 1/9 — CHHI Phase
Corona Virus Infection (Infections and infestations) | 0/9 | 1/5 | 0 | 0/9 — CHHI Phase
Post Viral Fatigue Syndrome (Infections and infestations) | 0/9 | 1/5 | 0 | 0/9 — CHHI Phase
Urethritis (Infections and infestations) | 0/9 | 0/5 | 1 | 0/9 — CHHI Phase
Viral Infection (Infections and infestations) | 0/9 | 0/5 | 1 | 0/9 — CHHI Phase
Gastroenteritis (Infections and infestations) | 0/9 | 0/5 | 0 | 1/9 — CHHI Phase
Syphilis (Infections and infestations) | 0/9 | 0/5 | 0 | 1/9 — CHHI Phase
Vulvovaginal Mycotic Infection (Infections and infestations) | 0/9 | 0/5 | 0 | 2/9 — CHHI Phase
Sunburn (Injury, poisoning and procedural complications) | 1/9 | 0/5 | 0 | 0/9 — CHHI Phase
Muscle Strain (Injury, poisoning and procedural complications) | 0/9 | 1/5 | 1 | 0/9 — CHHI Phase
Arthropod Bite (Injury, poisoning and procedural complications) | 0/9 | 0/5 | 1 | 0/9 — CHHI Phase
Contusion (Injury, poisoning and procedural complications) | 0/9 | 0/5 | 1 | 1/9 — CHHI Phase
Skin Abrasion (Injury, poisoning and procedural complications) | 0/9 | 0/5 | 2 | 0/9 — CHHI Phase
Thermal Burn (Injury, poisoning and procedural complications) | 0/9 | 0/5 | 1 | 0/9 — CHHI Phase
Alanine Aminotransferase Increased (Investigations) | 1/9 | 0/5 | 0 | 0/9 — CHHI Phase
Blood Pressure Systolic Increased (Investigations) | 2/9 | 0/5 | 0 | 0/9 — CHHI Phase
Eosinophil Count Increased (Investigations) | 8/9 | 2/5 | 10 | 8/9 — CHHI Phase
White Blood Cell Count Increased (Investigations) | 2/9 | 1/5 | 4 | 4/9 — CHHI Phase
Blood Pressure Diastolic Increased (Investigations) | 0/9 | 1/5 | 2 | 0/9 — CHHI Phase
Haemoglobin Decreased (Investigations) | 0/9 | 3/5 | 0 | 0/9 — CHHI Phase
Blood Pressure Increased (Investigations) | 0/9 | 0/5 | 1 | 0/9 — CHHI Phase
Fluid Retention (Metabolism and nutrition disorders) | 1/9 | 0/5 | 0 | 0/9 — CHHI Phase
Back pain (Metabolism and nutrition disorders) | 1/9 | 0/5 | 0 | 0/9 — CHHI Phase
Arthralgia (Metabolism and nutrition disorders) | 0/9 | 0/5 | 0 | 2/9 — CHHI Phase
Headache (Nervous system disorders) | 2/9 | 0/5 | 6 | 6/9 — CHHI Phase
Dizziness (Nervous system disorders) | 0/9 | 0/5 | 0 | 1/9 — CHHI Phase
Depression (Psychiatric disorders) | 0/9 | 0/5 | 1 | 0/9 — CHHI Phase
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1/9 | 0/5 | 0 | 4/9 — CHHI Phase
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0/9 | 0/5 | 0 | 2/9 — CHHI Phase
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0/9 | 0/5 | 0 | 3/9 — CHHI Phase
Upper-airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0/9 | 0/5 | 0 | 2/9 — CHHI Phase
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1/9 | 1/5 | 0 | 0/9 — CHHI Phase
Ecchymosis (Skin and subcutaneous tissue disorders) | 2/9 | 0/5 | 1 | 1/9 — CHHI Phase
Pruritus (Skin and subcutaneous tissue disorders) | 3/9 | 0/5 | 3 | 6/9 — CHHI Phase
Rash (Skin and subcutaneous tissue disorders) | 1/9 | 0/5 | 0 | 2/9 — CHHI Phase
Rash Macular (Skin and subcutaneous tissue disorders) | 0/9 | 0/5 | 1 | 0/9 — CHHI Phase
Injection Site Pain (General disorders) | 10 | 7 | 8 | 6
Injection Site Tenderness (General disorders) | 10 | 8 | 10 | 6
Injection Site Erythema (General disorders) | 1 | 1 | 2 | 0
Injection Site Swelling (General disorders) | 1 | 2 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 4 | 8 | 2 | 8
Nausea (Gastrointestinal disorders) | 0 | 4 | 2 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 5 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1 | 1
Application Site Pain (General disorders) | 0/9 | 0/5 | 2 | 1/9 — CHHI Phase
Application Site Tenderness (General disorders) | 1/9 | 0/5 | 2 | 2/9 — CHHI Phase
Application Site Rash (General disorders) | 7/9 | 2/5 | 4 | 4/9 — CHHI Phase
Application Site Swelling (General disorders) | 3/9 | 1/5 | 4 | 3/9 — CHHI Phase
Application Site Pruritus (General disorders) | 5/9 | 5/5 | 5 | 4/9 — CHHI Phase
Abdominal Pain (Gastrointestinal disorders) | 4/9 | 3/5 | 6 | 5/9 — CHHI Phase
Abdominal Bloating (Gastrointestinal disorders) | 5/9 | 3/5 | 6 | 5/9 — CHHI Phase
Nausea (Gastrointestinal disorders) | 4/9 | 3/5 | 6 | 6/9 — CHHI Phase
Vomiting (Gastrointestinal disorders) | 2/9 | 1/5 | 1 | 3/9 — CHHI Phase
Diarrhoea (Gastrointestinal disorders) | 3/9 | 1/5 | 6 | 4/9 — CHHI Phase
Flatulence (Gastrointestinal disorders) | 5/9 | 1/5 | 7 | 6/9 — CHHI Phase
Cough (Respiratory, thoracic and mediastinal disorders) | 4/9 | 0/5 | 1 | 4/9 — CHHI Phase
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2/9 | 2/5 | 1 | 4/9 — CHHI Phase

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-10-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT03172975/Prot_002.pdf
  • Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT03172975/SAP_001.pdf